CLINICAL TRIAL: NCT06804512
Title: Intermittent Visual Perturbations to Enhance Balance Training
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB202302204; 2R01NS104772-06A1 (NIH)
Record Dates: First submitted 2025-01-21; First posted 2025-02-03 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Balance
Keywords: walking balance; gait

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of 9 different training conditions. The intervention is walking on a treadmill mounted balance beam while wearing goggles that can perturb vision intermittently.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Control - No Goggles (Placebo Comparator): Participants will complete the balance beam walking practice without any changes to vision.
  Interventions: Device: Visual Occlusion Goggles; Behavioral: Balance Beam Walking
- Intervention - Goggles Worn But Turned Off (Experimental): Participants will complete the balance beam walking practice while wearing the goggles, but they will not be turned on.
  Interventions: Device: Visual Occlusion Goggles; Behavioral: Balance Beam Walking
- Intervention - Vision for 3.75s and Occlusion for 1.5s (Experimental): Participants will complete the balance beam walking practice while wearing the goggles. Vision time will be set to 3.75s, and the occlusion time will be set to 1.5s for the duration of the practice time.
  Interventions: Device: Visual Occlusion Goggles; Behavioral: Balance Beam Walking
- Intervention - Vision for 7.5s and Occlusion for 0.75s (Experimental): Participants will complete the balance beam walking practice while wearing the goggles. Vision time will be set to 7.5s, and the occlusion time will be set to 0.75s for the duration of the practice time.
  Interventions: Device: Visual Occlusion Goggles; Behavioral: Balance Beam Walking
- Intervention - Vision for 7.5s and Occlusion for 1.5s (Experimental): Participants will complete the balance beam walking practice while wearing the goggles. Vision time will be set to 7.5s, and the occlusion time will be set to 1.5s for the duration of the practice time.
  Interventions: Device: Visual Occlusion Goggles; Behavioral: Balance Beam Walking
- Intervention - Vision for 7.5s and Occlusion for 3s (Experimental): Participants will complete the balance beam walking practice while wearing the goggles. Vision time will be set to 7.5s, and the occlusion time will be set to 3s for the duration of the practice time.
  Interventions: Device: Visual Occlusion Goggles; Behavioral: Balance Beam Walking
- Intervention - Vision for 15s and Occlusion for 1.5s (Experimental): Participants will complete the balance beam walking practice while wearing the goggles. Vision time will be set to 15s, and the occlusion time will be set to 1.5s for the duration of the practice time.
  Interventions: Device: Visual Occlusion Goggles; Behavioral: Balance Beam Walking
- Intervention - Low Visible Light Transmission (Experimental): Participants will complete the balance beam walking practice while wearing the goggles. Vision time will be set to 7.5s, and the occlusion time will be set to 1.5s for the duration of the practice time. The visible light transmission will be set to a low value around 20% instead of total blackout for the occlusion time.
  Interventions: Device: Visual Occlusion Goggles; Behavioral: Balance Beam Walking
- Intervention - High Visible Light Transmission (Experimental): Participants will complete the balance beam walking practice while wearing the goggles. Vision time will be set to 7.5s, and the occlusion time will be set to 1.5s for the duration of the practice time. The visible light transmission will be set to a high value around 90% instead of total blackout for the occlusion time.
  Interventions: Device: Visual Occlusion Goggles; Behavioral: Balance Beam Walking

INTERVENTIONS:
Device: Visual Occlusion Goggles — The visual occlusion goggles alternate between sight and visual occlusion in a regular and programmable pattern. Based on the electrical properties of the goggles, they are also able to have the tint adjusted instead of blacking out entirely for the occlusion times during the programmed timings.
  Other Names: Senaptec
Behavioral: Balance Beam Walking — Participants will walk on a treadmill mounted balance beam to assess their balance

SUMMARY:
The purpose of this research study is to determine if intermittent visual perturbations can improve balance training. The investigators will quantify differences in body movement, muscle activity, and beam walking performance during and after practice walking on a balance beam that is 1" high. The investigators will ask the participants to come to the laboratory twice (2 sessions). The first session will not last more than 3 hours. The second session will not last more than 1 hour and will be two weeks after the first session. In total, the maximum amount of time the participant would be asked to participate is 4 hours.

DETAILED DESCRIPTION:
The investigators will recruit both younger (18-30 years of age) and older (65-89 years of age) participants. Half of the subjects will be male and half will be female. All subjects will walk on a treadmill-mounted beam for training and testing with a width determined by the challenge point approach. The beam width will vary for all participants based on the functional abilities of each individual.

When all subjects are consented into the study, the participant will walk across 6 different beams with differing widths laid on the ground. After practicing each width five times, the participant will start on the widest beam (7.6 cm) and walk across it three times. If the participant manages to reach the end of the beam (~3 m) without stepping off, that is a successful traverse. If the participant steps off the beam, it is not a successful traverse. The participant will either proceed to the next beam in the progression or stop at that beam width. That is the participant's starting beam width for the first training session. During the training session, if the participant goes 5 minutes without stepping off the beam, the investigators will move down to the next size beam to increase the participant's challenge level.

All the participants will wear liquid crystal lens goggles (Senaptec) during training. The goggles are sold commercially. The investigators can vary the length of time for unrestricted vision and for occluded vision.

Participants will be randomly assigned to different conditions that vary the parameters of brief intermittent visual perturbations provided by the goggles. One control group will not wear the goggles and one control group will wear the goggles but have no perturbations to their vision. Other groups will have varying lengths of occlusions and/or varying lengths of unobstructed vision. Another two groups will have different levels of light transmission in the goggles intermittently.

Subjects will come to the laboratory twice for training and testing. The first visit will be a pre-test, 30 minutes of training, and a post-test, Two weeks later, the participant will come back for one post-test. For both sessions, participants will wear motion analysis markers, inertial measurement sensors, and electromyography sensors on their body. For pre-tests and post-tests, participants will walk on the treadmill-mounted beam for 5 minutes without wearing the goggles. For training, they will complete three, 10-minute practice sessions walking on the beam for a total of 30 minutes of practice. The speed of the treadmill will be 0.22 m/s. The 30 minutes of training will be broken down into three 10-minute bouts with 5 minutes of rest in between. After completing the training on the first day, subjects will rest for 15 minutes and then complete a 5-minute post-test without the goggles. In the second day of testing 2 weeks later, participants will return to the lab to complete a 5-minute retention test of walking on the balance beam to measure step off errors. During beam walking on the treadmill, subjects will wear a safety harness about their torso that is connected to an overhead support to protect against falls.

Investigators will also assess cross-transfer of the beam walking training, with and without intermittent visual occlusions, to a secondary balance metrics. Participants will complete a single leg stance test before the beam walking pre-test and on the day of retention testing. Subjects will be asked to stand quietly with eyes open while the investigators monitor the time they are able to stand on one leg. Subjects will stand barefoot on the limb of their choice, with the other limb raised so that the raised foot is near but not touching the ankle of their stance limb. Each subject will be asked to focus on a spot on the wall at eye level in front with their vision. Subjects will cross their arms over the chest. Investigators will use a stopwatch to measure the amount of time the subject can stand on one limb. Time will commence when subjects raise their foot off the floor. Time will end when the subject either: (1) uncrossed arms, (2) moved the raised foot, (3) moved the weight-bearing foot to maintain balance, OR (4) 45 seconds elapses. The procedure will be repeated 3 times.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-30 years, or 65-89 years.
* Ability to walk independently for 10 minutes continuously.
* Willingness to be randomized to any experimental group and to participate in all aspects of study assessment and intervention

Exclusion Criteria:

-Major cognitive disorder that interferes with independence, based on affirmative response (always/usually/sometimes) to the following question: "As a result of confusion or memory loss, how often do you need assistance with day-to-day activities such as cooking, cleaning, taking medications, driving, or paying bills? Would you say it is 1) Always; 2) Usually; 3) Sometimes; 4) Rarely; or 5) Never".

* Current or recent (within 6 months) lower limb musculoskeletal injury that causes pain during walking or limits walking ability.
* History of neurological injury or disability (including spinal cord injury, stroke, Parkinson's disease, or multiple sclerosis).
* Difficulty communicating with study personnel.
* Current enrollment in any other clinical trial.
* Low vision that cannot be corrected by wearing contact lens. Low vision will be operationally defined as visual acuity less than 20/70 on standard eye chart, or difficulty perform complex walking tasks due to visual conditions affecting accurate navigation around and over obstacles (self-reported or observed by examiner). The goggles to be used in the study do not permit eyeglasses while using them.
* Illiterate or non-English speaking, due to the likelihood of difficulties following protocol instructions.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Balance Changes Between Pre and Post-Tests | Each subject completes the study in two weeks
  The primary outcome is a change in balance between the pre-test and post-tests and the pretest and follow-up. For the pre-test, post-test, and follow-up, participants will walk on the treadmill-mounted beam for 5 minutes without wearing the goggles. The pre-test will occur before the training periods begin, the post-test will occur after the training periods, and the follow-up occurs two weeks after the the first training. Step offs and time on the beam is recorded for each trial to make balance comparisons. The step offs and time on the beam used in conjunction to get step offs per minute by dividing step offs by time on the beam. Balance will be measured in step offs per minute.

SECONDARY OUTCOMES:
Balance Changes Between Static, Single Leg Standing on the Day of Training and Follow-up | Each subject completes the study in two weeks
  The secondary outcome will be a change in balance of the single legged balance between the first day and follow-up. Subjects will be asked to stand quietly with eyes open, standing barefoot on the limb of their choice, with the other limb raised so that the raised foot is near but not touching the ankle of their stance limb, looking forward, and with their arms crossed over their chest. This will be done any beam walking is done on both days. The subjects will be timed, ending when they uncross their arms, move their raised foot, move their weight bearing foot, or 45 seconds elapse. This will be done three times on each day. The times will then be compared between the first day of training and the follow-up to look for improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
We are currently not planning on publishing in an ICMJE journal.